CLINICAL TRIAL: NCT03356509
Title: The Effect of a High Intensity Interval Exercise Bout on Addictive Behaviors in Overweight/Obese Adults
Brief Title: Effect of Exercise on Chocolate Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Arlette Perry, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20170895
Record Dates: First submitted 2017-10-25; First posted 2017-11-29 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Acute Exercise and Addictive Behavior
MeSH Terms: conditions — Behavior, Addictive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): They will do a 26-min bout of high intensity interval exercise.
  Interventions: Behavioral: Exercise
- No exercise (No Intervention): They will sit quietly for 26 minutes without access to electronic devices or reading materials.

INTERVENTIONS:
Behavioral: Exercise — Exercise will be performed on a stationary bicycle ergometer.
  Arms: Exercise

SUMMARY:
The study will use stress inducing tasks to determine if there are significant improvements in mood, chocolate cravings, and attentional bias to chocolate in overweight/obese chocolate abusers following rest and a bout of high intensity interval exercise.

DETAILED DESCRIPTION:
The purpose of this research study is to investigate whether a single high intensity interval exercise (HIIE) bout, following two stress-inducing tasks, reduces addictive behavior to chocolate. Volunteers must complete the consent form before being able to participate in two days of testing (exercise day and control day) which will be presented in randomized order. The two days will be separated by a one to 7 day washout period. Subjects will be required to submit a three day chocolate diary then abstain from chocolate on the 4th day. They will also be asked to record everything they eat and drink on the day before and the morning of the study and list three types of chocolate they crave most. Two stress-inducing tasks will be performed on both days followed by completion of either 26 minutes of HIIE or seated resting condition followed by the completion of two mood and craving questionnaires. They will finally be asked to complete a task that measures the amount of attention they pay to chocolate. Statistical analyses will be conducted to determine the effect of either exercising or not on addictive behaviors to chocolate.

ELIGIBILITY:
Inclusion Criteria:

* BMI equal or greater than 25
* Eat at least 3.5 oz of chocolate per day
* Scorer at least 33 out of a possible 36 on the Handedness Questionnaire
* Ability to provide informed consent
* No medical contraindications to exercise
* Premenopausal

Exclusion Criteria:

* PMS
* Pregnancy
* Prisoners
* Risk factors for heart disease as determined by physician
* Medication that interferes with capacity to exercise
* Answer "Yes" to PAR-Q

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Attentional Bias (AB) to chocolate using a modified visual dot probe task (Kemps et al, 2009) | 15 minutes
  AB will be measured using a modified visual dot probe task, which consists of measuring reaction times to neutral images versus chocolate images (Kemps et al, 2009). Neutral images will consist of non-chocolate related items (i.e. office supplies). After 5 practice trials, 60 critical trials will be displayed which consist of either chocolate or neutral images (presented side by side). A black fixation cross will appear behind one of the images, and the subject has to respond as quickly as possible to which image the cross is located behind. The faster the subject responds to the cross behind the chocolate image, the higher their attentional bias is to chocolate. AB will be measured on both days following both the exercise and control conditions.

SECONDARY OUTCOMES:
Affective Valence measured by The Feeling Scale (Hardy & Rejeski, 1989) | 1 minute
  The Feeling Scale measures affective valence using an 11 point range from -5 to +5 with higher values indicating more pleasure. It is administered on both days following both the exercise and the control condition.
Affective Activation measured by the Felt Arousal Scale (Svebak & Murgatroyd, 1985) | 1 minute
  The Felt Arousal Scale measures affective activation using a 6 point range from 1 to 6 with the higher values indicating greater activation and arousal. It is administered on both days following both the exercise and the control condition.
Cravings for chocolate using the State Food Cravings Questionnaire (Cepeda-Benito et al, 2000) | 5 minutes
  This questionnaire measures the acute intensity of chocolate cravings using 15 items with 3 items per dimension. The five state dimensions of food cravings are: an intense desire to consume food, anticipation of positive reinforcement from eating, anticipation of relief from negative states and feelings as a result of eating, lack of control over eating if food is eaten, and craving as a hunger/physiological state. The dimensions will be evaluated using a 5 point Likert scale with the higher score meaning more intense cravings for chocolate. The questionnaire will be administered on both days following both the exercise and the control condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Clinical and Applied Physiology, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No